CLINICAL TRIAL: NCT06836193
Title: Do Emotions and Pain Combined Affect Mechanical Pain Thresholds and Other Pain-related Variables in Individuals with Chronic Pain
Brief Title: Do Emotions Affect Mechanical Pain Thresholds in Individuals with Chronic Pain?
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Linnaeus University (Other)
Responsible Party: Principal Investigator, Helena Gunnarsson, Dr, Linnaeus University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Dnr 2024-07781-01
Record Dates: First submitted 2025-02-12; First posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: PRESSURE PAIN THRESHOLD
Keywords: Pressure Pain Threshold; Pain; Emotion
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Negative emotional condition (Experimental): The participant will watch a short video-clip with negative emotional content.
  Interventions: Other: Emotional intervention
- Positive emotional condition (Experimental): The participant will watch a short video-clip with positive emotional content.
  Interventions: Other: Emotional intervention
- Neutral emotional condition (Sham Comparator): The participant will watch a short video-clip with neutral emotional content.
  Interventions: Other: Emotional intervention
- No emotional condition (Sham Comparator): The participant will wait for 2.30 minutes without any instructions about how to engage their thoughts.
  Interventions: Other: Emotional intervention

INTERVENTIONS:
Other: Emotional intervention — Negative emotional intervention
  Arms: Negative emotional condition; Neutral emotional condition
Other: Emotional intervention — Positive emotional intervention
  Arms: No emotional condition; Positive emotional condition

SUMMARY:
The purpose of this study is to investigate if different emotional states could influence mechanical pain thresholds in individuals with chronic pain.

DETAILED DESCRIPTION:
Participants will be randomized into 4 different groups watching different short video-clips (2.20 min). The negative emotions group will watch an uncomfortable short video containing violence and blood, the positive emotions group will watch a video containing a stand-up comedy show, the neutral emotions group will watch a video about how to paint a house, and the control group will just wait for 2.20 min, without any instructions about what to think about. Pressure pain thresholds will be measured with an algometer before and after the video-clips.

ELIGIBILITY:
Inclusion criteria

* Above 18 years of age
* Fluent in Swedish
* Persistent chronic pain with duration > 6 months Exclusion criteria
* Known neurological disease

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Pressure pain thresholds will be measured in kPa | The measurement takes place at the intervention session. First a baseline measurement is conducted, then comes the intervention and then the intervention measurement takes place.
  Pressure pain thresholds will be measured in kPa using a handheld algometer (Somedic AB).

IPD SHARING:
Plan to Share IPD: Undecided